CLINICAL TRIAL: NCT01359176
Title: The Capnography Library: Data Collection From Healthy Participants
Brief Title: Capnography Data Collection From Healthy Participants
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D0006376C
Record Dates: First submitted 2011-05-16; First posted 2011-05-24 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers

SUMMARY:
Capnography is the non-invasive monitoring of the concentration or partial pressure of carbon dioxide (CO2) in the expired respiratory gases; it is thus a non-invasive monitoring technique which allows fast and reliable insight into ventilation, circulation and metabolism. The capnogram is a direct monitor of the inhaled and exhaled concentration or partial pressure of CO2, and an indirect monitor of the CO2 partial pressure in the arterial blood. The purpose of this study is to create a waveform library by collecting CO2 waveform data from healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the trial by volunteer themself or by their legal guardian

Exclusion Criteria:

* Any individual who does not consent themselves or their legal guardian does not grant consent to participate in the trial
* A medical history of heart disease, lung disease, smoking, hypertension, pregnancy, diabetes or any other illness that excludes the participant from enrolling in the trial in the opinion of the PI

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To gather data received from monitoring healthy participants as reference for the creation of a capnography waveform library. | One hour
  Participants will put on the capnography monitoring device (a simple tube with prongs that fit in the nostrils, similar in design to the oxygen delivering device "nasal cannula") and this device will be hooked up to a computer. The participants will be asked to do very simple activities, such as sit, stand, eat and drink. The changes in their CO2 waveforms during these activities will be recorded in order to build a library of reference waveforms.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Einav, MD, Principal Investigator — Shaare Zedek Medical Centre
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel